CLINICAL TRIAL: NCT05809375
Title: Investigation of the Effects of a Client-centered Coping Skills Training in Individuals With Migraine: A Randomized Controlled Study
Brief Title: Coping Skills Training in Individuals With Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Etkin Bagi, Msc Occupational Therapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HU-ERG-EB-01
Record Dates: First submitted 2023-03-22; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Migraine
Keywords: Migraine; Pain; Coping Skills; Quality of Life
MeSH Terms: conditions — Migraine Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This study was designed as an assessor-blind, randomized controlled, and parallel-group study.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be performed by an investigator who was blinded to group allocation. Coping Skills Training was given to the control group participants, if they wanted to, after the final evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coping Skills Training Group (Active Comparator): Coping skills training (CST) will be given to the intervention group in line with the goals of the International Headache Society. Of the participants included in this study, the ones in the intervention group will be evaluated before and after the intervention.
  Interventions: Other: Coping Skills Training
- Control Grup (No Intervention): The participants in the control group will be evaluated at the beginning and after four weeks. CST will be given to the control group participants, if they want to, after the final evaluation.

INTERVENTIONS:
Other: Coping Skills Training — In the intervention, it was acted in a way to include the educational content determined by the International Headache Association and with a problem-solving perspective. The coping skills training contents in the literature were combined, and the CST prepared by including the most used and related contents will be given. CST includes a targeted therapy specifically developed for this study to address the needs and expectations of individuals with migraine. The targeted CST was designed by the authors, consisting of an occupational therapist, and two physiotherapists with clinical, and academic experience. It is planned as a total of eight sessions, and two sessions per week. CST includes giving information about migraine, activity tempo, progressive muscle relaxation exercise, stress management, social participation, leisure time management, general evaluation of the program, and home program.
  Arms: Coping Skills Training Group

SUMMARY:
This study was planned to investigate the effects of coping skills training on pain, quality of life, disability level, and coping skills in individuals with migraine.

DETAILED DESCRIPTION:
Migraine is a type of headache that lasts 4-72 hours, and it is characterized by throbbing pain on one side of the head, and recurrent attacks, making routine daily activities and movements difficult. Also, nausea and vomiting may accompany migraine, and sensitivity to both light and sound may increase. The World Health Organization (WHO) lists migraine as the disease that causes the most disability.

Approaches to the treatment of migraine consist of pharmacological and non-pharmacological treatments. Within the scope of non-pharmacological approaches, it is aimed to increase the coping skills of the individual by using methods such as exercise, stress management, and cognitive behavioral therapy, which include physical, mental, and cognitive interventions. Although these approaches are effective respectively, since migraine affects the whole life of the individual, there is a need for applications in which the approaches are applied with a combined and individual perspective. It has been shown that coping skills training improves both the physical and mental health and well-being of individuals with chronic headaches. It is known to cause a decrease in pain intensity, migraine attacks, and drug use. At the same time, it is aimed to adapt the individual to live efficiently. Despite these positive effects, there is a limited number of studies examining the effect of migraine coping skills training on individuals' disabilities and coping skills. Therefore, within the scope of this study, the effects of client-centered coping skills training on pain, disability, coping skills, and quality of life were examined.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of migraine meeting the International Headache Society diagnostic criteria (ICHD-3 beta International Classification of Headache Disorders),
* to be between the ages of 18-65,
* to have a migraine onset age younger than 50 (migraine onset age shouldn't be 50 years or more because being above is usually a secondary reason)
* to be literate.

Exclusion Criteria:

* have psychotic disorders, organic brain damage, other types of headaches, a history of traumatic head injuries, neck pain, any pathology causing headaches in the head and neck,
* alcohol or substance use,
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | four weeks
  The patients are asked to rate the average pain perception they felt during the day in a 10 cm straight line. The beginning of the line means "0 = no pain," and the end of the line means "10 = maximal pain."

SECONDARY OUTCOMES:
Nottingham Health Profile (NHP) | four weeks
  The Quality of life of the participants is assessed by using the NHP. It consists of 38 items assessing how severe an impact the respondent thinks their health is having on six dimensions: sleep, physical mobility, energy, pain, emotional reactions, and social isolation. Every item has a different weight, depending on the severity of the symptom. The sum of the weighted scores is 100 for each subdimension. Thus, summing all weighted values of every item, the score between 0 and 100 is obtained for each subdimension. The total score was obtained by summing the scores of six subdimensions, giving values between 0 and 600. Higher scores indicate a greater level of distress. The NHP is valid and reliable in Turkish populations.
Migraine Disability Assessment Score (MIDAS) | four weeks
  It consists of five questions that measures the influence of headaches on three domains of activity over the preceding 3 months: paid and school work, household work, and leisure activities with family or in social situations. MIDAS measures the number of days in which migraine interferes with these activities, and establishes four disability grades: minimal, mild, moderate, and severe disability. The MIDAS is valid and reliable in Turkish populations.
The brief COPE | four weeks
  The Brief COPE measures strategies for coping with stress and includes 14 subscales in which two items are grouped into two coping strategies: effective approach coping (active coping, acceptance, positive reframing, planning, use of emotional or instrumental support) and ineffective avoidant coping (denial, self-distraction, substance use, behavioural disengagement, venting, and self-blame). Each question has a selection range from 1 ("I have not been doing this at all") to 4 ("I have been doing this a lot"), and the higher subscale scores indicate using those coping strategies more. The Brief COPE is valid and reliable in Turkish populations.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Ekici, Principal Investigator — Hacettepe University; Mahmut Yaran, Study Chair — Ondokuz Mayıs University

IPD SHARING:
Plan to Share IPD: No